CLINICAL TRIAL: NCT01959516
Title: Multicenter, Randomized, Blinded, Two-period Cross-over Study to Assess the Effect of Glycopyrronium (44 Micrograms QD) Versus Tiotropium (18 Micrograms QD) on Morning Symptoms and Pulmonary Function in Patients With Moderate to Severe COPD
Brief Title: Effect of Glycopyrronium on Morning Symptoms and Pulmonary Function in Patients With Moderate to Severe COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CNVA237A3401
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Results first posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-03

CONDITIONS: COPD
Keywords: COPD, early morning symptoms
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence A ⇒ B (Experimental): Participants will receive sequence A = glycopyrronium + placebo to tiotropium during 28 days, followed by a 14 day washout period, then sequence B= tiotropium + placebo to glycopyrronium for 28 days.
  Interventions: Drug: Glycopyrronium; Drug: Tiotropium; Drug: Placebo to glycopyrronium; Drug: Placebo to tiotropium
- Sequence B ⇒ A (Experimental): Participants will receive sequence B= tiotropium + placebo to glycopyrronium during 28 days, followed by a 14 day washout period, then sequence A= glycopyrronium + placebo to tiotropium for 28 days.
  Interventions: Drug: Glycopyrronium; Drug: Tiotropium; Drug: Placebo to glycopyrronium; Drug: Placebo to tiotropium

INTERVENTIONS:
Drug: Glycopyrronium — Glycopyrronium capsule for inhalation once per day via SDDPI
Drug: Tiotropium — Tiotropium capsule for inhalation once per day via HandiHaler® device
Drug: Placebo to glycopyrronium — Placebo to glycopyrronium capsule for inhalation once per day via SDDPI
Drug: Placebo to tiotropium — Placebo to tiotropium capsule for inhalation once per day via HandiHaler® device

SUMMARY:
This study purpose is to further study the profiles of glycopyrronium (NVA237) and tiotropium during the first hours after dosing and their impact on pulmonary function, COPD symptoms and ability to perform daily activities by the patient.

DETAILED DESCRIPTION:
Randomized, multicenter, blinded, two-period cross-over design. Each treatment will last 28 days. All patients will receive both treatments in a cross-over design, with a wash-out period of 14-19 days in between. The total duration of the study for each patient is approximately 70 days (from randomization) plus 30 days of safety follow-up.

ELIGIBILITY:
Inclusion criteria:

* Male and female adults aged ≥ 40 years.
* Co-operative outpatients with a clinical diagnosis of moderate to severe COPD confirmed by spirometry according to GOLD criteria 2013 and including all of the following: a) Current or ex-smokers who have a smoking history of at least 10 pack years (e.g.10 pack years = 1 pack /day x 10 years or ½ pack/day x 20 years). An ex-smoker may be defined as a subject who has not smoked for ≥ 6 months at Screening. b) Patients with airflow limitation indicated by a post-bronchodilator FEV1 < 80% and ≥ 40% of the predicted normal value at Visit 2 (Post- bronchodilator refers to within 10-15 min of inhalation of 400 µg (4x100 µg) of salbutamol). c) .Post-bronchodilator FEV1/FVC < 0.7 at Visit 2 (Post- bronchodilator refers to within 10-15 min of inhalation of 400 µg (4x100 µg) of salbutamol).
* Patients with a COPD Assessment Test (CAT) score ≥ 10 at Visit 2.

Exclusion criteria:

* Patients who have had a COPD exacerbation requiring systemic glucocorticosteroid treatment or antibiotics and/or hospitalization in the 6 weeks prior to Visit 1. In the event of an exacerbation occurring during the Screening period (Visits 1-2), the patient must be discontinued from the study. The patient may be re-enrolled once the inclusion/exclusion criteria are met. Only one re-enrollment is allowed.
* Patients who have had a respiratory tract infection within 6 weeks prior to Visit 1. Patients who develop a respiratory tract infection between Visit 1 and Visit 2 must discontinue from the trial, but may be permitted to re-enrol at a later date once the inclusion/exclusion criteria have been met. Only one re-enrollment is allowed.
* Patients on any long-acting bronchodilator therapy. Those patients may enter the study after bronchodilator withdrawal during a 10-day wash-out period (only rescue salbutamol allowed as bronchodilator therapy during wash-out). Patients on fixed combination of long acting β2-agonists/inhaled corticosteroid (LABA/ICS) therapy before screening must be switched to the equivalent dose of ICS monotherapy and salbutamol as rescue.
* Patients receiving any other prohibited COPD-related medications specified in Table 5-1 must undergo the required wash-out period prior to Visit 2.
* Patients who have had a clinical history of asthma.
* Patients with concomitant pulmonary disease, e.g. pulmonary tuberculosis or clinically significant bronchiectasis.
* Patients with alpha-1-antitrypsin deficiency.
* Patients with contraindications for LAMA treatment including medical history of symptomatic prostatic hypertrophy, bladder neck obstruction, narrow-angle glaucoma and severe renal impairment (estimated glomerular filtration rate below 30 ml/min/1.73 m2) documented in the previous 6 months.
* Patients with a history of unstable cardiovascular disease or arrhythmias including atrial fibrillation/flutter or long QT syndrome or whose resting QTcF (calculated according to Fridericia QT correction formula preferred, but Bazett acceptable) is prolonged (≥ 450 msec for males and ≥ 460 msec for females) at screening (Visit 1) or baseline (Visit 2, baseline 1).
* Concomitant use of agents known to prolong the QT interval unless it can be permanently discontinued for the duration of study.
* Patients contraindicated for treatment with, or having a history of reactions/ hypersensitivity to any of the following inhaled drugs, drugs of a similar class or any component thereof: -anticholinergic agents - long and short acting 2 agonists -sympathomimetic amines -excipients of the trial medication (lactose monohydrate and/or magnesium estearate)
* Patients whose body mass index (BMI) is less than 15 or greater than 40 kg/m2.
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.

Other exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2014-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (20):
- Germany (8):
  - Novartis Investigative Site, Berlin, Germany
  - Novartis Investigative Site, Potsdam, Germany
  - Novartis Investigative Site, Wiesbaden, Germany
  - Novartis Investigative Site, Geesthacht, Schleswig-Holstein
  - Novartis Investigative Site, Berlin, State of Berlin
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Leipzig
- Italy (3):
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Orbassano, TO
- Spain (3):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Lugo, Galicia
  - Novartis Investigative Site, Zaragoza, Zaragoza
- United Kingdom (6):
  - Novartis Investigative Site, Cambridge, United KIngdom
  - Novartis Investigative Site, Watford, United Kingdom
  - Novartis Investigative Site, Blackpool
  - Novartis Investigative Site, Bradford
  - Novartis Investigative Site, Cardiff
  - Novartis Investigative Site, Wishaw

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 126 patients were randomized to one of the two treatment sequences in a ratio of 1:1. Due to misrandomization, two patients did not receive at least one dose of the study treatment. Both, safety and ITT population included 124 patients.
Groups:
- Glycopyrronium First, Then Tiotropium": Sequence A (Glycopyrronium 44 μg QD+ placebo of tiotropiumto) to B (Tiotropium 18 μg QD + placebo of glycopyrronium) Sequence B (Tiotropium 18 μg QD + placebo of glycopyrronium) to A (Glycopyrronium 44 μg QD+ placebo of tiotropiumto)
- Tiotropium First, Then Glycopyrronium: Sequence B (Tiotropium 18 μg QD + placebo of glycopyrronium) to A (Glycopyrronium 44 μg QD + placebo of tiotropiumto) Sequence A (Glycopyrronium 44 μg QD+ placebo of tiotropiumto) to B (Tiotropium 18 μg QD + placebo of glycopyrronium)
Period: Epoch 1
Arm/Group | Glycopyrronium First, Then Tiotropium" | Tiotropium First, Then Glycopyrronium
Started | 63 | 63
Safety Population | 62 | 62
ITT Population | 62 | 62
Completed | 53 | 58
Not Completed | 10 | 5
Not completed — Adverse Event | 4 | 1
Not completed — unsatisfactory therapeutic effect | 1 | 0
Not completed — Subject withdrew consent | 3 | 2
Not completed — Administrative problems | 1 | 0
Not completed — Use of prohibited treatment | 1 | 0
Not completed — Moderate or severe COPD exacerbation | 0 | 1
Not completed — Protocol deviation | 0 | 1
Period: Epoch 2
Arm/Group | Glycopyrronium First, Then Tiotropium" | Tiotropium First, Then Glycopyrronium
Started | 63 | 63
Completed | 61 | 62
Not Completed | 2 | 1
Not completed — unsatisfactory therapeutic effect | 1 | 0
Not completed — Subject withdrew consent | 1 | 0
Not completed — Moderate or severe COPD exacerbation | 0 | 1

BASELINE CHARACTERISTICS:
Population: The intention-to-treat (ITT) population consisted of all randomized patients who received at least one dose of the study treatment and had at least one post-dose value of FEV1
Groups:
- All Participants (Intent To Treat Analysis,ITT): All participants who were randomized to one of the two treatment sequences in a ratio of 1:1. Participants will receive sequence A = glycopyrronium + placebo to tiotropium during 28 days, followed by a 14 day washout period, then sequence B= tiotropium + placebo to glycopyrronium for 28 days.
Arm/Group | All Participants (Intent To Treat Analysis,ITT)
Number analyzed (Participants) | 124
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.7 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 87

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in 1 Second (FEV1) AUC0-4h After First Dose of Treatment.
Description: Forced Expiratory Volume in 1 second (FEV1) Area Under the Curve (AUC) will measured via spirometry and calculated from 0 to 4 hours post-dose on day 1 of study treatment.
Time Frame: Day 1
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters*hours
Groups:
- Glycopyronium From Sequence A to B and Sequence B to A: Sequence A (Glycopyrronium 44 μg QD+ placebo of tiotropiumto) to B (Tiotropium 18 μg QD + placebo of glycopyrronium) Sequence B (Tiotropium 18 μg QD + placebo of glycopyrronium) to A (Glycopyrronium 44 μg QD+ placebo of tiotropiumto)
- Tiotropium From Sequence A to B and Sequence B to A: Sequence B (Tiotropium 18 μg QD + placebo of glycopyrronium) to A (Glycopyrronium 44 μg QD + placebo of tiotropiumto) Sequence A (Glycopyrronium 44 μg QD+ placebo of tiotropiumto) to B (Tiotropium 18 μg QD + placebo of glycopyrronium)
Arm/Group | Glycopyronium From Sequence A to B and Sequence B to A | Tiotropium From Sequence A to B and Sequence B to A
Number analyzed (Participants) | 124 | 124
Liters*hours | 1.7432 (0.5171) [1.7132 to 1.7732] | 1.7132 (0.5175) [1.6830 to 1.7434]
Statistical Analysis 1: Comparison: Glycopyronium From Sequence A to B and Sequence B to A vs Tiotropium From Sequence A to B and Sequence B to A; Test type: Superiority or Other; p = 0.0250, Mixed Models Analysis

2. Secondary Outcome: Comparison of Glycopyrronium QD Versus Tiotropium QD on Symptoms Outcome
Description: Comparison of symptoms outcome between glycopyrronium QD versus tiotropium QD will be conducted via the PROMorning COPD Symptoms questionnaire. This questionnaire will be completed by participants at waking-up, pre-inhalation of study treatment (at home), and they will complete Part 2 of PRO-Morning COPD Symptoms questionnaire at site, 3hours post-inhalation of study treatment. The PRO-Morning COPD Symptoms Questionnaire is a self-administered patient reported outcome (PRO) instrument developed by the sponsor to evaluate patients' experience of early morning symptoms of COPD. The questionnaire consists of two parts : predose and postdose.
  Each part has 6 questions and for each question a scale of 0 to 10 can be reached. For the predose and postdose part of the questionnaire you will have then each a total score of 0-60 by adding the sub-scores for each question, higher scores represent worse severity of COPD morning symptoms
Time Frame: day 1 (baseline) and week 4
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Glycopyronium From Sequence A to B and Sequence B to A | Tiotropium From Sequence A to B and Sequence B to A
Number analyzed (Participants) | 124 | 124
Scores on a scale
  3h post-dose (Day 1) | 9.7068 (8.8) [8.7294 to 10.6841] | 10.3974 (8.1) [9.4036 to 11.3913]
  3h post-dose (Week 4) | 10.4641 (8.8) [9.3786 to 11.5496] | 10.3193 (9.3) [9.2286 to 11.4100]
Statistical Analysis 1: Comparison: Glycopyronium From Sequence A to B and Sequence B to A vs Tiotropium From Sequence A to B and Sequence B to A; Test type: Superiority or Other; p = 0.1439, Mixed Models Analysis

ADVERSE EVENTS:
Arm/Group | Glycopyronium From Sequence A to B and Sequence B to A | Tiotropium From Sequence A to B and Sequence B to A
Serious Adverse Events (participants affected / at risk) | 2/124 | 2/124
Other Adverse Events (participants affected / at risk) | 17/124 | 12/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Glycopyronium From Sequence A to B and Sequence B to A (N=124) | Tiotropium From Sequence A to B and Sequence B to A (N=124)
Pneumonia (Infections and infestations) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Glycopyronium From Sequence A to B and Sequence B to A (N=124) | Tiotropium From Sequence A to B and Sequence B to A (N=124)
Bundle branch block left (Cardiac disorders) | 1 | 0
Bundle branch block right (Cardiac disorders) | 1 | 0
Cystoid macular oedema (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Hepatic cyst (Hepatobiliary disorders) | 0 | 1
Food allergy (Immune system disorders) | 1 | 0
Dermatophytosis (Infections and infestations) | 1 | 0
Infected dermal cyst (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 3 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Presyncope (Nervous system disorders) | 1 | 1
Sciatica (Nervous system disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Balanoposthitis (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety